CLINICAL TRIAL: NCT04497025
Title: Feasibility and Safety of an Immersive Virtual Reality-based Vestibular Rehabilitation Program for Dizziness, Balance and Fatigue Improvement in People With Multiple Sclerosis: Protocol for a Pilot Randomised Controlled Study
Brief Title: Conventional Vestibular Training Versus Immersive Virtual Reality- Based Vestibular in Multiple Sclerosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maria Jesus Casuso-Holgado (Other)
Responsible Party: Sponsor-Investigator, Maria Jesus Casuso-Holgado, Assistant Professor, University of Seville
Organization: University of Seville (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RVEM2020
Record Dates: First submitted 2020-07-18; First posted 2020-08-04 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Multiple Sclerosis; Vestibular Disease; Dizziness; Balance Disorders; Fatigue; Quality of Life; Usability; Cybersickness
MeSH Terms: conditions — Multiple Sclerosis; Vestibular Diseases; Dizziness; Fatigue

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immersive virtual reality-based vestibular training. (Experimental): Subjects in this group will receive the same intervention than the other group of study, but they will wear a 3D head mounted display (Oculus Quest glasses) and will receive real-time gaming feedback in terms of visual and audio output while using the training system.
  Participants will receive a total of 20 sessions (3 sessions of 50 minutes per week, 7 weeks). These sessions will be divided in 10 initial sessions (based on the three first blocks of Cawthorne-Cooksey protocol) and 10 advanced sessions in which vestibular exercises are gradually get more complicated by modifiying the following exercise parameters: base of support width, standing on unstable surface, alternatives single leg support, tandem position, increased velocity of head movements, higher head range motion and coordinated movements with arms and trunk.
  Same location, tailoring parameters and physical therapist supervision than conventional vestibular training.
  Interventions: Other: Immersive Virtual-based vestibular rehabilitation
- Conventional vestibular training. (Active Comparator): Subjects in the control group will receive a total of 20 sessions of 50 minutes (3 sessions per week, 7 weeks). They will receive traditional "Cawthorne-Cooksey" vestibular rehabilitation exercises. This program improves vestibular compensation through a mechanism of neuroplasticity known as adaptation, habituation and substitution. Just like the virtual reality intervention it will be divided in 10 initial sessions and 10 advanced sessions. For the advanced phase of intervention exercises parameters were the same described for the virtual vestibular rehabilitation intervention.
  A physical therapy with at least two years of expertise in vestibular rehabilitation will adjust the difficulty level. The intervention will be conducted at the Physical Therapy Department of the University of Sevilla (Spain).
  Interventions: Other: Conventional vestibular rehabilitation protocol

INTERVENTIONS:
Other: Immersive Virtual-based vestibular rehabilitation — Vestibular rehabilitation based on virtual environment using a head mounted display
  Arms: Immersive virtual reality-based vestibular training.
Other: Conventional vestibular rehabilitation protocol — "Cawthorne-Cooksey" vestibular rehabilitation exercises.
  Arms: Conventional vestibular training.

SUMMARY:
The effectiveness of convectional vestibular training for balance and dizziness rehabilitation in people with multiple sclerosis has been recently demonstrated in a meta-analysis by this research team (doi: 10.3390/jcm9020590). Furthermore, non-immersive virtual reality-based environments seem to be useful for balance and gait rehabilitation in this population (doi: 10.1177/0269215518768084). However, nothing is known about the feasibility and effectiveness of immersive virtual reality-based rehabilitation in people with multiple sclerosis.

The primary aim of this research is to determine the feasibility, safety and effectiveness of an immersive virtual reality-based vestibular training for dizziness, balance and fatigue rehabilitation, compared to conventional vestibular training.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female subjects from 18-65 years old
* Clinically diagnosed with any type of multiple sclerosis in accordance with the revised McDonald criteria
* With walking ability according to the Expanded Disability Status Scale score (EDSS =6)
* With the objective presence of dizziness symptoms (Dizziness Handicap Inventory = 16)

Exclusion Criteria:

* Blurred vision
* Cognitive impairment (Mini Mental State Examination =24)
* Another neurologic disorder contributing to balance impairment
* Relapse within the last 3 months
* Changes in pharmacotherapy within the last 3 months
* History of vestibular rehabilitation within the last 6 months
* Acute cardiovascular of respiratory illness
* Any other contraindication to physical activity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of virtual reality-based vestibular rehabilitation | 7 weeks of intervention
  Usability of virtual reality device: System Usability Scale (0-100%). Higher Scores means higher usability
  Participation rate
  Retention rate
  Adherence to treatment rate
Safety of virtual reality-based vestibular rehabilitation | 7 weeks of intervention
  Cybersickness: Scores ranging between 10 and 15 mean significant symptoms and above 20 indicates a simulator problem
  Falls registry
  Adverse events registry

SECONDARY OUTCOMES:
Change from baseline dizziness symptoms at 7 weeks | 7 weeks after intervention
  Dizziness Handicap Inventory (0-100 points). Higher scores mean worse dizziness symptoms.
Change from baseline static balance at 7 weeks | 7 weeks after intervention
  Static balance assessed by posturography Dynamic balance assessed by Balance Berg Scale. Higher score better balance.
Change from baseline fatigue at 7 weeks | 7 weeks after intervention
  Modified Fatigue Impact Scale (0-84 points). Higher scores mean worse fatigue symptoms.
Change from baseline quality of life at 7 weeks | 7 weeks after intervention
  Multiple Sclerosis Quality of Life Scale 54 (0-100 points). Higher values indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Jesus Casuso-Holgado, Principal Investigator — University of Seville
Locations (1):
- Universidad de Sevilla, Seville, Spain

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR

REFERENCES:
- [Derived] Garcia-Munoz C, Casuso-Holgado MJ, Hernandez-Rodriguez JC, Pinero-Pinto E, Palomo-Carrion R, Cortes-Vega MD. Feasibility and safety of an immersive virtual reality-based vestibular rehabilitation programme in people with multiple sclerosis experiencing vestibular impairment: a protocol for a pilot randomised controlled trial. BMJ Open. 2021 Nov 22;11(11):e051478. doi: 10.1136/bmjopen-2021-051478. PMID 34810187